CLINICAL TRIAL: NCT03991494
Title: A Phase 1 Study to Investigate the Absorption, Metabolism, and Excretion of [14C]Pamiparib Following Single Oral Dose Administration in Patients With Advanced and/or Metastatic Solid Tumors
Brief Title: Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-Pamiparib in Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BGB-290-106; 2018-001156-36 (EudraCT Number)
Record Dates: First submitted 2019-06-14; First posted 2019-06-19 (Actual); Results first posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pamiparib (Experimental)
  Interventions: Drug: [14C]-pamiparib

INTERVENTIONS:
Drug: [14C]-pamiparib — During the treatment phase, pamiparib 60 mg administered orally twice daily

SUMMARY:
This is an open-label study, in participants with advanced and/or metastatic solid tumors, which consists of 2 parts: a research phase (inpatient) and a treatment phase. The research phase (Part 1) of the study will assess the disposition of a single oral dose of [14C]-pamiparib. In the treatment phase (Part 2) participants will be allowed to have continued access to pamiparib.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically and/or cytologically confirmed advanced or metastatic solid tumor that has progressed after treatment with approved therapies for which there are no standard therapies available
2. A total body weight between 50 and 100 kg, inclusive at Screening
3. Measurable disease by CT/MRI
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
5. Adequate organ function

Key Exclusion Criteria:

1. Clinically significant cardiovascular disease
2. Have a previous complete gastric resection, chronic diarrhea, active inflammatory gastrointestinal disease, or any other disease causing malabsorption syndrome.
3. Poor peripheral venous access
4. Major surgical procedure, open biopsy, or significant traumatic injury ≤ 2 weeks prior to Day 1, or anticipation of need for major surgical procedure during the course of the study
5. Use or have anticipated need for food or drugs known to be strong or moderate CYP3A inhibitors or strong CYP3A inducers

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2020-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (2):
- United Kingdom (2):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - Royal Liverpool University Hospital Clinical Research Unit, Liverpool

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Mu S, Palmer D, Fitzgerald R, Andreu-Vieyra C, Zhang H, Tang Z, Su D, Sahasranaman S. Human Mass Balance and Metabolite Profiling of [14 C]-Pamiparib, a Poly (ADP-Ribose) Polymerase Inhibitor, in Patients With Advanced Cancer. Clin Pharmacol Drug Dev. 2021 Sep;10(9):1108-1120. doi: 10.1002/cpdd.943. Epub 2021 Apr 19. PMID 33876576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 2 parts: a Research Phase (Part 1) in which participants were inpatients and a Treatment Phase (Part 2) in which participants were outpatients.
Pre-assignment Details: Potential participants were screened to assess their eligibility to enter the study within 28 days prior to administration of the first dose. Up to 10 participants could be enrolled to ensure that 4 participants completed Part 1 of the study.
Groups:
- Pamiparib: Research Phase (Part 1): participants received a single dose of 60 mg [14C]-pamiparib orally Treatment phase (Part 2): participants received pamiparib 60 mg twice daily orally
Period: Overall Study
Arm/Group | Pamiparib
Started | 4
Completed | 0
Not Completed | 4
Not completed — Progressive Disease | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4

OUTCOME MEASURES:

1. Primary Outcome: Plasma Pamiparib Pharmacokinetics: Area Under the Concentration-time Curve (AUC) From Time Zero to Infinity (AUC0-∞)
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliLiter (h*ng/mL)
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
hours*nanograms/milliLiter (h*ng/mL) | 29300 (21.6)

2. Primary Outcome: Plasma Total Radioactivity and Whole Blood Total Radioactivity Pharmacokinetics: AUC From Time Zero to Infinity (AUC0-∞)
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received at least on dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ngEq/g
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
h*ngEq/g
  Plasma Total Radioactivity | 42200 (21.5)
  Whole Blood Total Radioactivity | 32200 (16.2)

3. Primary Outcome: Plasma Pamiparib Pharmacokinetics: AUC From Time Zero to the Last Quantifiable Concentration (AUC0-t)
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received at least on dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
h*ng/mL | 29200 (21.6)

4. Primary Outcome: Plasma Total Radioactivity and Whole Blood Total Radioactivity Pharmacokinetics: AUC From Time Zero to the Last Quantifiable Concentration (AUC-t)
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received at least on dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ngEq/g
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
h*ngEq/g
  Plasma Total Radioactivity | 41800 (21.6)
  Whole Blood Total Radioactivity | 31200 (16.1)

5. Primary Outcome: Plasma Pamiparib Pharmacokinetics: Maximum Observed Concentration (Cmax) of Pamiparib
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received at least on dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
ng/mL | 2190 (12.4)

6. Primary Outcome: Plasma Total Radioactivity and Whole Blood Total Radioactivity Pharmacokinetics: Maximum Observed Concentration (Cmax)
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received at least on dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/g
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
ngEq/g
  Plasma Total Radioactivity | 2390 (9.0)
  Whole Blood Total Radioactivity | 1730 (11.8)

7. Primary Outcome: Plasma Pamiparib Pharmacokinetics: Time of Cmax (Tmax)
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received at least on dose of [14C]-pamiparib and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
hours | 2.00 [1.00 to 3.05]

8. Primary Outcome: Plasma Total Radioactivity Whole Blood Total Radioactivity Pharmacokinetics: Time of Cmax (Tmax)
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received at least on dose of [14C]-pamiparib and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
hours
  Plasma Total Radioactivity | 2.25 [1.50 to 3.05]
  Whole Blood Total Radioactivity | 2.25 [1.50 to 3.05]

9. Primary Outcome: Plasma Pamiparib Pharmacokinetics: Apparent Terminal Elimination Half-Life (t1/2)
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
hours | 29.2 (6.02)

10. Primary Outcome: Plasma Total Radioactivity and Whole Blood Total Radioactivity Pharmacokinetics: Apparent Terminal Elimination Half-Life (t1/2)
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
hours
  Plasma Total Radioactivity | 21.6 (10.3)
  Whole Blood Total Radioactivity | 13.3 (3.13)

11. Primary Outcome: Plasma Pamiparib Pharmacokinetics: Apparent Total Clearance (CL/F)
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (L/h)
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
Liters/hour (L/h) | 2.21 (23.2)

12. Primary Outcome: Plasma Pamiparib Pharmacokinetics: Apparent Volume of Distribution (Vz/F)
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
Liters | 91.3 (18.5)

13. Primary Outcome: Plasma Pamiparib Pharmacokinetics: AUC0-∞ of Plasma Pamiparib Relative to AUC0-∞ of Plasma Total Radioactivity
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received at least on dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Groups:
- Pamiparib: Research Phase (Part 1): participants received 60 mg [14C]-pamiparib twice daily orally
  Treatment phase (Part 2): participants received pamiparib 60 mg twice daily orally
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
Ratio | 0.694 (2.7)

14. Primary Outcome: Plasma Pharmacokinetics: AUC0-∞ of Whole Blood Total Radioactivity to AUC0-∞ of Plasma Total Radioactivity
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 6, 12, 24, 48, 72, 96, 120, and 144 hours post-dose on Day 1 to Day 7
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
Ratio | 0.764 (5.8)

15. Primary Outcome: Percentage of Total Radioactivity Excreted in Urine
Time Frame: 192 hours of [14C]-Pamiparib Administration
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: % Excreted
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
% Excreted | 57.84 (5.12)

16. Primary Outcome: Cumulative Urinary Excretion of Pamiparib
Time Frame: 192 hours of [14C]-Pamiparib Administration
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
mg | 1.095 (40.2)

17. Primary Outcome: Renal Clearance of Pamiparib (CLR)
Time Frame: 192 hours of [14C]-Pamiparib Administration
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: CLR (L/h)
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
CLR (L/h) | 0.03742 (59.5)

18. Primary Outcome: Fecal Recovery of Total Radioactivity
Time Frame: 192 hours of [14C]-Pamiparib Administration
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: % Excreted
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
% Excreted | 26.89 (6.83)

19. Primary Outcome: Cumulative Recovery of Total Radioactivity in Total Excreta
Time Frame: 192 hours of [14C]-Pamiparib Administration
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: % Excreted
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
% Excreted | 84.73 (3.53)

20. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events in Part1 and Part 2
Time Frame: Up to 6 months
Population: The safety population for Part 1 consisted of all participants who received 1 dose of study drug, 60 mg [14C]-pamiparib in Part 1 and the safety population for Part 2 consisted of all participants who participated in Part 1 and received at least 1 dose of 60 mg pamiparib in Part 2.
Measure: Number; unit: number of participants
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
number of participants
  Part 1: Number of Participants with AEs | 4
  Part 1: Participants with SAEs | 0
  Part 2: Number of Participants with AEs | 3
  Part 2: Participants with SAEs | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Time Frame: Up to 6 months
Population: The safety population for Part 1 consisted of all participants who received 1 dose of study drug, 60 mg [14C]-pamiparib, in Part 1 and the safety population for Part 2 consisted of all participants who participated in Part 1 and received at least 1 dose of 60 mg pamiparib in Part 2.
Measure: Number; unit: number of participants
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
number of participants | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in 12-lead ECG Parameters, Vital Signs Data, Physical Examinations and Weight Data
Time Frame: Up to 6 months
Population: The safety population for Part 1 consisted of all participants who received at least 1 dose of study drug, 60 mg [14C]-pamiparib, in Part 1 and the safety population for Part 2 consisted of all participants who participated in Part 1 and received at least 1 dose of 60 mg pamiparib in Part 2.
Measure: Number; unit: Number of participants
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
Number of participants | 0

23. Secondary Outcome: Pamiparib Metabolite Identified and Metabolic Profile Using Measured Mass (M3)
Description: Human plasma, urine, and feces samples were analyzed by LC-MS.
Time Frame: 0.5, 1, 2, 6, 12, 24, 48, 72, 96, 120, and 144 hours post dose on Days 1 to 7
Population: The PK population included all participants who received one dose of [14C]-pamiparib and had evaluable PK data.
Measure: Number; unit: Da
Arm/Group | Pamiparib
Number analyzed (Participants) | 4
Da | 313.1098

ADVERSE EVENTS:
Time Frame: Approximately 30 days after the last dose of pamiparib - up to 6 months
Groups:
- Pamiparib: Research Phase (Part 1): participants received a single dose of 60 mg [14C]-pamiparib orally Treatment phase (Part 2): participants received 60 mg pamiparib twice daily orally
Arm/Group | Pamiparib
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pamiparib (N=4)
Constipation (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Amylase increased (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Headache (Nervous system disorders) | 1
Influenza like illness (General disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Oedema peripheral (General disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Sinusitis (Infections and infestations) | 1
Tremor (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT03991494/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT03991494/SAP_001.pdf